CLINICAL TRIAL: NCT02456675
Title: A Phase 2, Open-Label Study of the Safety and Efficacy of INCB40093 and INCB40093 Combined With Itacitinib (INCB039110) in Subjects With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: INCB040093 and INCB040093 Combined With Itacitinib (INCB039110) in Relapsed/Refractory Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision was made to terminate the study due to the changing treatment landscape for the development of new agents in combination in Hodgkin lymphoma.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40093-201
Record Dates: First submitted 2015-03-19; First posted 2015-05-28 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Refractory Hodgkin Lymphoma; Recurrent Adult Hodgkin's Lymphoma
Keywords: Refractory Hodgkin lymphoma; Relapsed Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INCB040093 Monotherapy (Experimental): INCB040093 sustained release (SR) tablets will be administered orally twice daily (BID) without regard to food.
  Interventions: Drug: INCB040093 Monotherapy
- INCB040093 and itacitinib (INCB039110) Combination Therapy (Experimental): Subjects allocated to Group B will be given INCB040093 BID in combination with itacitinib SR tablets. The dose of itacitinib will be orally given once daily (QD). Doses should be taken in the morning on an empty stomach if possible.
  Interventions: Drug: INCB040093; Drug: itacitinib

INTERVENTIONS:
Drug: INCB040093 Monotherapy — INCB040093 sustained release (SR) tablets will be administered orally twice daily (BID) without regard to food.
  Arms: INCB040093 Monotherapy
Drug: INCB040093 — INCB040093 sustained release (SR) tablets will be administered orally twice daily (BID) without regard to food.
  Arms: INCB040093 and itacitinib (INCB039110) Combination Therapy
Drug: itacitinib — The dose of itacitinib will be given orally once daily (QD).
  Other Names: INCB039110
  Arms: INCB040093 and itacitinib (INCB039110) Combination Therapy

SUMMARY:
A Phase 2, open-label study to evaluate the safety and efficacy of INCB040093 as monotherapy and as combination therapy with itacitinib (INCB039110) in subjects with relapsed or refractory Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years or older
* Histologically confirmed diagnosis of classical HL
* Must be relapsed or refractory after autologous stem cell transplant (ASCT) and/or 2 or more prior chemotherapy regimens
* Must have had prior treatment with brentuximab vedotin or not a candidate for treatment with brentuximab vedotin
* Eastern Cooperative Oncology Group (ECOG) 0 to 2

Exclusion Criteria:

* Laboratory parameters not within the protocol-defined range
* Received an investigational study drug within 28 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study drug.
* Received any approved anticancer medications within 21 days or 5 half-lives (whichever is longer) prior to receiving their first dose of study drug EXCEPT steroids at ≤ 10 mg prednisone daily (or equivalent).
* Has any unresolved toxicity ≥ Grade 2 from previous anticancer therapy
* Received autologous stem cell transplant within 28 days or allogeneic transplant within 3 months prior to first dose of study drug
* History of lymphoma involving the central nervous system
* Evidence of active or prior hepatitis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as determined by the percentage of subjects achieving a partial response (PR) or complete response (CR) | Measured every 9 weeks from baseline until progression (estimated to be 12 months)
  Evaluate the efficacy of INCB040093 as monotherapy and when given in combination with itacitinib by assessing the objective response rate (ORR) determined by an independent review committee.

SECONDARY OUTCOMES:
Percentage of participants reporting adverse events in the monotherapy group | every 3 weeks for the duration of participation in the study [estimated to be 12 months]
  Safety and tolerability of INCB040093 as monotherapy in subjects with relapsed or refractory Hodgkin's lymphoma (HL) as determined by clinical laboratory assessments, physical exams, 12-lead ECG and summary of adverse events
Percentage of participants reporting adverse events in the combination therapy group | every 3 weeks for the duration of participation in the study [estimated to be 12 months]
  Safety and tolerability of INCB040093 when given in combination with itacitinib in subjects with relapsed or refractory Hodgkin's lymphoma (HL) as determined by clinical laboratory assessments, physical exams, 12-lead ECG and summary of adverse events
Percentage of subjects achieving a complete response (CR) determined by the independent review committee and based on standard response criteria | Week 36 disease evaluation
  Complete Response is determined by the independent review committee and based on standard response criteria defined by the Response Evaluation Criteria in Solid Tumor (RECIST) criteria. CR: Disappearance of all target and nontarget lesions.
To evaluate the duration of response (DOR) | Week 36 disease evaluation
  Duration of response is defined as the time from the first assessment showing response (CR or PR) determined by the independent review committee to the first documented disease progression determined by the independent review committee or death due to any cause, whichever occurs first.
To evaluate the progression-free survival (PFS) | Week 36 disease evaluation
  PFS was defined as the time from first dose to the first documented disease progression or relapse as assessed by independent review committee or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation